CLINICAL TRIAL: NCT05441345
Title: Sarcopenia and Short Bowel Syndrome: the Microbiota-gut-muscle Axis
Brief Title: Sarcopenia and Short Bowel Syndrome
Acronym: SARCO-SGC
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220496
Record Dates: First submitted 2022-06-17; First posted 2022-07-01 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Short Bowel Syndrome
Keywords: Sarcopenia; short bowel syndrome; adaptation
MeSH Terms: conditions — Short Bowel Syndrome; Sarcopenia | interventions — Surveys and Questionnaires; Urination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SBS patients
  Interventions: Other: questionnaires with collection of stool and urine

INTERVENTIONS:
Other: questionnaires with collection of stool and urine — questionnaires will be completed (GPAQ, SarQoL, EQ-5D-3L, SF36), with collection of stool (for care and research) and urine

SUMMARY:
Sarcopenia or the loss of skeletal muscle is highly prevalent in many diseases, including short bowel syndrome (SBS). While adaptation is more likely in SBS patients with a colon-in-continuity, the consequences and underlying mechanisms are unclear. An overabundance of fecal Lactobacillus was found but not yet linked to adaptation or sarcopenia. The objectives are to study the evolution of sarcopenia and the link with intestinal adaptation in SBS.

DETAILED DESCRIPTION:
Patients with short bowel syndrome (SBS) will be screened and included in longitudinal or cross-sectional studies if eligible.

The longitudinal study will follow patients with type 1 SBS (enterostomy) before and every 3 months after continuity surgery for 1 year. Cross-sectional studies will follow patients with type 2 or 3 SBS (jejunocolonic or -ileal anastomosis) for 1 year (every 3 months during the first 2 years after continuity surgery or every 6 months after).

Study visits will include clinical examination, nutritional assessment, endoscopy with biopsies and/or intestinal absorption assessment planned as part of routine follow-up. In addition, questionnaires will be completed (GPAQ, SarQoL, EQ-5D -3L, SF36), with collection of stool (for routine and research) and urine samples (for research).

The objective are to study the evolution of sarcopenia and the link with intestinal adaptation in SBS. The results may identify metabolic or microbial biomarkers and predictors of nutritional optimisation in SBS, which is a complex and costly orphan disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* SBS diagnosis validated by small bowel length and either type 1 (enterostomy), type 2 or 3 (jejuno-colic or -ileal anastomosis)
* Patient not objecting to the collection of personal data as part of the study

Exclusion Criteria:

* Pregnancy

  * Remaining hail length unknown
  * Patient expressing opposition to participating in the cohort
  * Patients who are unable to express themselves

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients in CMS cared for and followed in the gastroenterology and nutritional assistance department of Beaujon Hospital
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2024-07-16 (Actual)

PRIMARY OUTCOMES:
Evolution of sarcopenia | at 12 months
  Changes in muscle strength (Jamar's dynamometer)
Evolution of sarcopenia | at 12 months
  Changes in muscle mass (bioimpedance analysis)

SECONDARY OUTCOMES:
Impact of sarcopenia | at 12 months
  Changes in questionnaire of quality of life SarQoL
Impact of sarcopenia | at 12 months
  Changes in questionnaire of quality of life EQ-5D-3L
Impact of sarcopenia | at 12 months
  Changes in questionnaire of quality of life SF36
Impact of sarcopenia | at 12 months
  Changes in questionnaire of physical activity (GPAQ)
Link with intestinal adaptation | at 12 months
  Number of changes in histological markers of adaptation in relation to sarcopenia. Each of these elements can be considered as a chang : crypt depths, villi length, immune cells.
Link with intestinal adaptation | at 12 months
  Changes in biological markers of adaptation in relation to sarcopenia: ApoB48, citrulline, leptin, nutrients
Quantification of intestinal adsorption and its link with intestinal adaptation | at 12 months
  Changes in intestinal absorption balance markers of adaptation in relation to sarcopenia: digestive losses in fat, proteins, carbohydrates and total energy. These elements will be quantified by biological assessements.
Link with intestinal adaptation | at 12 months
  Changes in bacterial fermentation markers of adaptation in relation to sarcopenia: D-lactate, short-chain fatty acids (SCFAs)
Quantification of urinary metabolite linked with sarcopenia | at 12 months
  Changes in urinary markers of fermentation in relation to sarcopenia (metagenomic sequencing)
Quantification of fecal metabolite linked with sarcopenia | at 12 months
  Changes in fecal markers of fermentation in relation to sarcopenia (mass spectrometry)

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie KAPEL, MPharma PhD, Principal Investigator — APHP
Locations (1):
- Service de Coprologie Fonctionnelle Hôpital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No